CLINICAL TRIAL: NCT03897920
Title: Doppler Ultrasound Renal Arterial Resistive Indices As Predictor Of Multiorgan Failure In Patients With Acute Hypoxic Respiratory Failure Admitted To Respiratory Intensive Care Unit (Cryptic Shock Index CSI- RICU)
Brief Title: Doppler Ultrasound Renal Arterial Resistive Indices As Predictor Of Multiorgan Failure In Patients With Acute Hypoxic Respiratory Failure Admitted To Respiratory Intensive Care Unit (Cryptic Shock Index- RICU)
Acronym: CSI-RICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Alessandro Marchioni, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio 6
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Failure; Multi Organ Failure
MeSH Terms: conditions — Respiratory Insufficiency; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Doppler ultrasound assessment of renal arteria resistive index — A high frequency probe will be used together with the use of color or power Doppler to help vessel localization. As resistance to blood flow progressively increases from the hilar arteries toward the more peripheral parenchymal vessels, renal arteria resistive index (RRI) will be done at the level of the arcuate or interlobar arteries, adjacent to medullary pyramids. Measurements will be repeated in different parts of both organs (superior, median, and lower) when at least three reproducible waveforms have been obtained. An RRI will be calculated with the following formula: (peak systolic velocity - end diastolic velocity)/peak systolic velocity, and the mean value of three measurements at each kidney is usually considered. An RRI value 0.60 ± 0.01 (mean ± SD) is usually taken as normal with a value of 0.70 being considered the upper normal threshold

SUMMARY:
Patients with de novo respiratory failure undergoing non invasive ventilation (NIV) present failure rates of mechanical ventilation ranging from 4 to 50%. Causes for NIV treatment failure are various but the onset of septic shock and subsequent multi-organ failure (MOF) seem play a critical role. Recent data show that the 37% of patients admitted to intensive care unit for de novo respiratory failure without any other organ failure experience multiple organ failure within the first days from admission. Early identification of hypoxic patients at major risk for MOF seems critical. Physiological studies have demonstrated that the underlying mechanisms for organ damage preceding MOF are those involved in the oxygen consumption (VO2)/oxygen delivery (DO2) mismatch. Doppler ultrasound indices of renal arteria resistance are directly correlated tot he VO2/DO2 mismatch. With this study we aim at investigating the correlation between Doppler ultrasound indices of renal arteria resistance in patients with de novo respiratory failure admitted to ICU and the onset of MOF within the first 7 days form admission.

ELIGIBILITY:
Inclusion Criteria:

* patients with de novo respiratory failure admitted to the respiratory intensive care unit of the university hospital of Modena

Exclusion Criteria:

* age lower than 18 or higher than 85
* presence of organ failure apart form lung failure at the time of admission in the respiratory intensive care unit
* pregnancy
* difficult or unreliable ultrasound window for renal arterial resistive index assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with de novo respiratory failure admitted to the respiratory intensive care unit of the university hospital of Modena without any other organ failure
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Onset of shock | 7 days from Respiratory Intensive Care Unit admission
  Shock will be clinically identified by a vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L (>18 mg/dL) in the absence of hypovolemia

IPD SHARING:
Plan to Share IPD: Undecided